CLINICAL TRIAL: NCT04269603
Title: Normal Values and Quality Assessment of Light Transmission Aggregometry (LTA) Using Aggregometer TA-8V (Stago®)
Brief Title: LTA Assessement Using Aggregometer TA-8V (Stago®)
Acronym: NORMAGREG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL19_0661
Record Dates: First submitted 2019-12-23; First posted 2020-02-17 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteer
Keywords: light transmission aggregometry; platelets; platelet functions; von Willebrand disease; quality assessment
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 30 healthy adult volunteers (Other): Healthy adult volunteers without hemorrhagic diathesis.
  Interventions: Device: Take blood (TA-8V (Stago®)

INTERVENTIONS:
Device: Take blood (TA-8V (Stago®) — Healthy volunteers will have 3 blood samples at M0, M3 and M6.

SUMMARY:
Exploring platelet functions requires aggregation tests platelet. The Haematology Laboratory of Hospices Civils de Lyon currently has two new TA-8V plate aggregation automatons® (Stago).

The supplier of these devices does not offer reference values for these tests. There are also no references in the data literature. Therefore reference values must be established from healthy volunteer subjects.

The use of these automatons is subject to the NF (French Standard) EN (European Standard) ISO (International Organization for Standardization) 15189 standard of the COFRAC ( French Accreditation Comity) that requires checking their proper functioning. This audit must be traced in a method validation folder.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged between 18 and 70 years
* Weighting more than 50 kg
* Subjects having signed informed consent
* Subjects registered in the French health-care system database

Exclusion Criteria:

* Personal history of anemia, thrombopenia, hemorrhagic disease
* Caffeine intake 2 hours prior to blood sampling
* Tobacco intake in the half hour prior to blood sampling
* Use of any drug impacting platelet function
* for antiplatelet agents: at least 10 days prior to blood sampling
* for anti-depressants: at least 10 days prior to blood sampling
* for non-steroid anti-inflammatories: at least 3 days prior to blood sampling
* Refusal to undergo the 3 visits and 3 blood samples of the study
* Refusal to sign the informed consent form
* No registration in the French Health-care system database
* Pregnant women and women who are breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Platelets aggregation results for LTA on TA-8V (Stago®) | Month 0
  Normal values for platelets aggregation will be established using various agonists to activate platelets. :
  • Ristocetin (STAGO®)
Platelets aggregation results for LTA on TA-8V (Stago®) | Month 3
  Normal values for platelets aggregation will be established using various agonists to activate platelets. :
  * Collagen (STAGO®)
  * ADP (adenosine diphosphate) (STAGO®)
  * Arachidonate (STAGO®)
  * TRAP (Thrombin Receptor Activating Platelet) (STAGO®)
Platelets aggregation results for LTA on TA-8V (Stago®) | Month 6
  Normal values for platelets aggregation will be established using various agonists to activate platelets. :
  * Epinephrine (STAGO®)
  * PMA (phorbol 12-myristate 13 acetate) (SIGMA®)
  * PAF (Platelet Activator Factor) (BACHEM®)
  * Ionophore calcium (SIGMA®)
  * 11-Epoxy (SIGMA®)
  * Prostaglandin E1 (SIGMA®)

SECONDARY OUTCOMES:
LTA intra assay variability | Month 0
  Intra assay variability of maximal platelet aggregation will be assessed by calculating a coefficient of variation of the studied parameters.
LTA intra assay variability | Month 3
  Intra assay variability of maximal platelet aggregation will be assessed by calculating a coefficient of variation of the studied parameters.
LTA intra assay variability | Month 6
  Intra assay variability of maximal platelet aggregation will be assessed by calculating a coefficient of variation of the studied parameters.
LTA inter operator variability | Month 0
  Inter operator variability of maximal platelet aggregation will be assessed by percentage of agreement (%).
LTA inter operator variability | Month 3
  Inter operator variability of maximal platelet aggregation will be assessed by percentage of agreement (%).
LTA inter operator variability | Month 6
  Inter operator variability of maximal platelet aggregation will be assessed by percentage of agreement (%).
Agonist reagents stability duration | up to 2 months post reagents reconstitution and 2 months post reconstitution with the same technician, the same automaton and the same healthy volunteer sample.
  Reagents will be reconstituted and stored at -20°C. They will be used for aggregation assay extemporaneously, 1 week, 2 weeks , 1 month and 2 months post reconstitution.
Agonist reagents stability duration | up to 2 months post reagents reconstitution
  Reagents will be reconstituted and stored at -20°C. They will be used for aggregation assay extemporaneously, 1 week, 2 weeks , 1 month and 2 months post reconstitution.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Haemostasis Unit/Haematology Laboratory, Groupement Hospitalier Est, Bron, France